CLINICAL TRIAL: NCT06741566
Title: Pre-operative Intra-nasal Dexmedetomidine or Insulin for Prevention of Early Post-operative Cognitive Dysfunction in Patients Undergoing Elective Coronary Artery Bypass Graft. A Comparative Randomized Bi-centric Study
Brief Title: Pre-operative Intra-nasal Dexmedetomidine or Insulin for Prevention of Early Post-operative Cognitive Dysfunction in Patients Undergoing Elective Coronary Artery Bypass Graft.
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, Ass professor anesthesia and pain, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 640/R
Record Dates: First submitted 2024-12-14; First posted 2024-12-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Post Operative Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator)
  Interventions: Drug: intranasal saline group
- Insulin group (Active Comparator)
  Interventions: Drug: intranasal insulin
- Dexmedetomidine group (Active Comparator)
  Interventions: Drug: Intranasal dexmedetomidine

INTERVENTIONS:
Drug: intranasal saline group — 3 ml of saline 0.9 % twice daily for 2 days preoperatively at fixed time ( 9 am and 6 pm)
  Arms: Control group
Drug: intranasal insulin — 20 IU of regular insulin on 3 ml saline 0.9% twice daily for 2 days preoperative via mucosal atomization device at fixed times ( 9 am, 6 pm)
  Arms: Insulin group
Drug: Intranasal dexmedetomidine — 1.5 mic/kg on 3 ml saline 0.9% twice daily for 2 days preoperative via mucosal atomization device at fixed times ( 9 am, 6 pm)
  Arms: Dexmedetomidine group

SUMMARY:
On pump coronary revascularization is a very common leading cause for post-operative cognitive dysfunction regarding patient age grouping and diffuse systemic inflammatory response induced by bypass machine . Many factors are incriminated as pre-operative sleep disturbance, previous history of neurocognitive dysfunction. The accumulating evidence refers to an incidence between 20-40% with majority among geriatric population. The primary pathology is still elusive and many trials are under evaluation. Neuro-inflammation, hypo perfusion, fat emboli and reperfusion injury are among the most postulative aetiologias. The corner stone in the pathology of postoperative cognitive dysfunction is abnormal sleep rhythm. Intra-nasal insulin can provide neuroprotection via providing insulin growth factor and obtund neuronal apoptosis , while dexmedetomidine can antagonize neural-degeneration via regulation of systematic inflammatory cytokines including interleukin 1β, tumor necrosis factor-α, and NF-κB, inhibiting the expressions of Toll-like receptor , and through α2 adrenoceptor-mediated anti-inflammatory pathways

ELIGIBILITY:
Inclusion Criteria:

* Adult population, 60 years or above, both sex, candidate for elective on pump coronary revascularization

Exclusion Criteria:

* Combined reperfusion and valve replacement operations.
* Emergency or redo CABG surgery.
* Preoperative MMSE less than 20
* Diabetic or chronic alcoholic population.
* Pre-operative cardiomyopathy (Ejection fraction less than 40%).
* Previous cerebro-vascular stroke or carotid endarterectomy.
* Previous history of carotid endarterectomy.
* History of heparin resistance.
* Preoperative history of dementia, language impairment, severe visual and hearing impairment, any psychiatric disorder.
* Chronic use of hynotics, mode stabilizing drugs or melatonin.
* Reoperation for emergency surgical issues during hospital stay.
* Patient refusal
* Loss to follow up ( patient dyscompliance, mortality)
* population with failed weaning from CPB and the use ventricular assisted device ( intraaortic ballon- impella)
* Pre or post operative pacing.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-27 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-05-11 (Estimated)

PRIMARY OUTCOMES:
Mini mental state examination | PREOPERATIVE, 1,3,5, days
  Acute cognitive assessment, score from 0-10 = severe sementia, 10-20 = moderate dementia, 20-25= mild , 25-30= questionably significabt

SECONDARY OUTCOMES:
Time for extubation | 6 hours
  hours elapsed from ICU admission until extubation
ICU stay | one week
  Days from ICU admission postoperative and discharge to word
serum glucose | 1 day before surgery, at time of surgery, at ICU admission, first day, second , third
  serum glucose
Serum troponin | preoperative, on admission, 3 days, 5 days
  normal level < 0.12
procedure related complication | 3 days
  bradycardia, spasm, cough,

OTHER OUTCOMES:
Pittsburgh Sleep Quality Index | preoperative assessment, score from 0-21. 0-10= very good sleep, 10-15= mild impairment, 15-21= significant sleep disturbance with higher score indicates poor sleep quality
  Patient sleep status in the last month
Richards-Campbell Sleep Questionnaire | preoperative, 1,3, 5, days postoperative
  sleep quality . The counting method was recorded with numbers (0 points to 100 points). The higher the score, the higher the sleep quality star.
Confusion assessment method - ICU | PREOPERTIVE, 1,3,5, DAYS
  POST PERATIVE DELERIUM. CAM includes four aspects: (1) acute onset and fluctuat- ing course, (2) inattention, (3) incoherent thinking, and (4) altered consciousness; the presence of both
  (1) and (2), and one of (3) or (4) is diagnostic of POD
  With a total score of 30, a higher score indicates a lower incidence of neurocognitive dysfunction
Epworth sleepiness scale | preoperative, 1,3,5 days after
  patient awarness of sleepiness. Eight questions each score from 0 to 3. 0-10= normal range.
  11-14=mild sleepiness.. 15-17= moderate sleepiness.... > 18= severe sleepiness
transcranial doppler | preoperative, 1 day, 3 days, 5 days
  Pulsatality index ( PI) > 0.8 means severe vasospasm
transcranial doppler | preoperative, 1 day, 3 days, 5 days
  resistive index .. 0.8> severe spasm